CLINICAL TRIAL: NCT05877495
Title: The Effect of Food Safety, Security and Waste Prevention Intervention on the Knowledge, Attitudes, Behavior and Practices (KAB-P) of University Students: A Randomized Controlled Trial
Brief Title: Food Safety, Security and Waste Prevention Intervention on the KAB-P Approach of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Nagihan Kırcali Haznedar, Research Assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22408003
Record Dates: First submitted 2023-03-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Educational Problems
Keywords: Food security; Food safety; Food waste; Nutrition education; Undergraduates; Sustainability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education Group (Experimental): The experimental group which is given the nutrition education about food security, safety and prevention food waste.
  First of all, a data collection form will be applied to the participants. This form contains food insecurity experience scale, food consumption frequency form, determination of waste level form, safety knowledge, attitudes and behaviors. The they will receive a 14-session training created by the researchers by examining the literature and various guides. This training includes about, prevention food waste with kitchen activities, food safety, food security and waste control. After this education participants will be answered the same questions again.
  Interventions: Behavioral: Nutritional Education Intervention
- Control Group (No Intervention): The control group will be asked the same data collection form with no intervention.
  After the post-tests the control group will be given the same education.

INTERVENTIONS:
Behavioral: Nutritional Education Intervention — A 14-session training created by the researchers by examining the literature and various guides. This training includes about, prevention food waste with kitchen activities, food safety, food security and waste control. The content of the intervention will be loaded soon.
  Arms: Nutrition Education Group

SUMMARY:
The goal of this clinical trial is aimed to examine the effect of food safety and security and waste reduction education on the knowledge, attitudes, behavior, and practices of undergraduates.

The main questions it aims to answer are:

Will the food consumption record of the experimental group be lower than the control group after the training? Will the experimental group's post-training food insecurity scale scores be higher than the control group? Will the experimental group's waste level be lower after the training than the control group? Will the experimental group's food safety knowledge test scores be higher than the control group?

DETAILED DESCRIPTION:
Initiatives aimed at ensuring access to safe, nutritious, and adequate food and the reduction of food waste are critical for social well-being and sustainable development. This project is aimed to examine the effect of food safety and security and waste reduction education on the knowledge, attitudes, behavior, and practices of undergraduates. The research was designed as a randomized controlled trial in which the pre-test-post-test method will be applied. The participants of the study will consist of 110 (n intervention = 55, n control = 55) students studying at Selcuk University with the G*Power 3.1.9.7 power analysis program. A grading randomization method will be used accordingly to the faculties. Through the research, participants will be provided with training consisting of 14 sessions on food safety, food security, and the reduction of food waste. Research data will be collected with; general information part, 24-hour recalled food consumption record, Food Insecurity Experience Scale, food consumption frequency form, management of food consumption-related behaviors, and food waste questionnaire form, and Food Safety, Attitudes, and Behaviors Scale. In addition, body weight (kg), height (m), waist (cm), hip (cm), and neck (cm) measurements will be taken from the participants in the study. The research findings will be analyzed by t-test in the groups dependent on the changes within the intervention and control groups; t-test in the independent groups. Furthermore, the Cohen d power level will be calculated, and the group time interaction between the groups will be evaluated by two-way analysis of variance and partial ETA recalculation in repetitive measurements. In case of data loss, a Little's Mcar test will be performed based upon the result of which the data will be analyzed and evaluated via the Intention-to-treat protocol by completing the data.

ELIGIBILITY:
Inclusion Criteria:University students who

* are not diagnosed with any chronic disease,
* do not use drugs constantly,
* do not follow a special diet,
* have not received any training on food safety-security and waste, and volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* diagnosed with chronic disease,
* use drug constantly,
* follow a special diet,
* received any training on food safety-security and waste

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Knowledge level | Baseline and week 14
  Comparison of mean scores between pre/post tests

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Aktas, Prof. Dr., Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)